CLINICAL TRIAL: NCT03160183
Title: Investigating Chemotherapy Treatments, Response and Subsets of HIV-associated Kaposi Sarcoma in Malawi
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC 1424
Record Dates: First submitted 2017-05-02; First posted 2017-05-19 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Kaposi Sarcoma; HIV
Keywords: initiating chemotherapy; prospective, open label, single arm, cohort; non randomized, non interventional
MeSH Terms: conditions — Sarcoma, Kaposi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify important associations between complete and comprehensive clinical, laboratory, and genomic data derived from patients and tumor specimens, with prospectively recorded clinical outcomes. The investigators also hope to move beyond simple risk factor associations as previously described, to develop a composite score specifically for KS recurrence or progression, analogous to widely used risk scores that are used to direct up-front treatment of other cancers. In so doing, the investigators will draw on extremely granular data to prospectively identify patients who are most likely to benefit from new treatments.

DETAILED DESCRIPTION:
This is a prospective, nonrandomized, open-label, single arm, cohort study of pathologically confirmed HIV-associated KS patients initiating chemotherapy in Malawi. The primary objective of this study is to estimate the complete response rate (CR by ACTG criteria) at 48 weeks. This will be done both overall and by chemotherapy (BV or not BV) treatment group. Secondary objectives are to estimate PFS and OS for both overall and by chemotherapy treatment group. Exploratory objectives include the investigation of: select clinical variables and laboratory biomarkers among HIV-associated KS patients and their possible association with response, PFS, and OS; the histopathology of KSHV-associated lymphoproliferative diseases among HIV-associated KS patients; KSHV strains in tumor biopsies, PBMC and plasma, and KSHV gene expression characteristics between KS that develops on and off ART.

The investigators plan to accrue 200 HIV-associated KS patients at a rate of approximately 50 patients per year. Approximately half of the patients will receive BV chemotherapy treatment. An important factor for this study's size is that it will be comparable to or exceed the size of other important KS cohort studies, which have demonstrated significant differences in outcomes based on gender or baseline KSHV DNA levels.

The investigators want to show that there are definable biologic and clinical subsets within the HIV-associated KS population, and that identifying these subsets will have direct relevance to more effective treatment strategies for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed KS initiating chemotherapy at Lighthouse Trust or the Kamuzu Central Hospital (KCH) Cancer Clinic
* HIV positive (confirmed at any time point prior by local standard of care assay) on or off ART
* Age ≥18 years
* Residence <200 kilometers from KCH
* Able to understand and comply with study procedures for the entire length of the study
* Subject able to understand and provide written consent in English or Chichewa Informed consent reviewed and signed by patient

Exclusion Criteria:

* Failure to meet inclusion criteria listed above.
* Specifically, pregnancy and breastfeeding are not exclusion criteria given the observational nature of the study with diagnostic and treatment interventions administered according to local standards of care.
* KS relapse disease as defined by a prior KS diagnosis within 1 year prior to enrollment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected adults ≥18 years of age with pathologically confirmed KS who are initiating chemotherapy at Lighthouse Trust or the KCH Cancer Clinic.
Sampling Method: Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2016-09; Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Estimate the complete response rate (CR) at 48 weeks of HIV-associated KS patients overall and by BV treatment group. | 48 weeks
  the assessment of a patient's response (CR) to chemotherapy at 48 weeks by ACTG criteria

SECONDARY OUTCOMES:
Estimate the Progression Free Survival (PFS) in HIV-associated KS patients overall and by bleomycin-vincristine (BV) treatment group | 48 weeks
  PFS which will be defined as the time from treatment initiation until disease progression or death
Estimate OS in HIV-associated KS patients overall and by BV treatment group | 48 weeks
  To estimate OS in HIV-associated KS patients overall and by BV treatment group

OTHER OUTCOMES:
The clinical variables and laboratory biomarkers among HIV-associated KS patients and their possible association with response, PFS, and OS | 48 weeks
  The prevalence and nature of lymphoproliferative diseases among HIV-associated KS patients
The histopathology of KSHV-associated lymphoproliferative diseases among HIV-associated KS patients | 48 weeks
  KSHV gene expression characteristics for HIV-associated KS that develops on and off antiretroviral therapy (ART)
The kind of KSHV strains in tumor biopsies, PBMC and plasma | 48 weeks
  Viral genome features of HIV-associated KS
The KSHV gene expression characteristics between KS that develops on and off ART | 48 weeks
  To describe KSHV gene expression characteristics between KS that develops on and off ART

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Dittmer, Principal Investigator — UNC-CH
Locations (2):
- Malawi (2):
  - UNC Project, Lighthouse Trust, Lilongwe
  - UNC Project, Lilongwe

IPD SHARING:
Plan to Share IPD: Undecided